CLINICAL TRIAL: NCT05443763
Title: Exploring the Experiences and Outcomes of a Summer Intensive Therapy Program- Mixed Methods Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jamie Hall, Assistant Teaching Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2090791
Record Dates: First submitted 2022-05-18; First posted 2022-07-05 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-06

CONDITIONS: Children With Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: Cohort study of children receiving intensive therapy and their caregivers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: An interdisciplinary intensive therapy program — Children will receive physical, occupation, and/or speech therapy 1-3 hours/day each for 4-5 days/week x 4 weeks.

SUMMARY:
The purpose of this study is to assess the effectiveness of an interdisciplinary intensive therapy program for ambulatory and non-ambulatory children with neurodevelopmental disorders across the ICF and to explore caregiver experiences and perspectives of the program.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effectiveness of an interdisciplinary intensive therapy program for ambulatory and non-ambulatory children with neurodevelopmental disorders across the ICF and to explore caregiver experiences and perspectives of the program. Research questions include: 1.) What are the effects of an intensive program on postural control and functional mobility for children with neurodevelopmental disorders? 2.) What are the effects of an intensive therapy program on dual tasking for children with neurodevelopmental disorders? 3.) What are the perceptions of caregivers of a multidisciplinary intensive therapy program for their children with neurodevelopmental disorders? Data will be gathered before and after the intensive program as part of usual care and ambulatory children will be further assessed in the motion analysis lab. Caregivers will complete a questionnaire about satisfaction with services and also a 4 question open-ended question survey about their experience with intensive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children receiving therapy through Children's Therapy Center's Tiger Intensive Program and their caregivers from May 23, 2022, to Aug 19, 2022.

Exclusion Criteria:

* none

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Instrumented Gait Analysis | before intensive therapy episode of care, approximately 4 weeks
  3D gait analysis in gait lab
Instrumented Gait Analysis | after intensive therapy episode of care, approximately 4 weeks
  3D gait analysis in gait lab
Center of pressure measure | after intensive therapy episode of care, approximately 4 weeks
  COP measure during balance task
Center of pressure measure | before intensive therapy episode of care, approximately 4 weeks
  COP measure during balance task
Measures of processes of care (MOPC) | after intensive therapy episode of care, an average of 4 weeks
  Questionnaire to assess satisfaction with therapy services
Timed up and go | before intensive therapy episode of care, an average of 4 weeks
  TUG assessment--timed assessment including standing from a chair, walking a distance and returning to the chair
Timed up and go | fter intensive therapy episode of care, an average of 4 weeks
  TUG assessment--timed assessment including standing from a chair, walking a distance and returning to the chair
Modified Clinical Test of Sensory Integration and Balance | after intensive therapy episode of care, an average of 4 weeks
  mCISIB--balance test in 4 conditions
Modified Clinical Test of Sensory Integration and Balance | before intensive therapy episode of care, an average of 4 weeks
  mCISIB--balance test in 4 conditions
Pediatric Balance Scale | before intensive therapy episode of care, an average of 4 weeks
  PBS-balance test
Pediatric Balance Scale | after intensive therapy episode of care, an average of 4 weeks
  PBS-balance test
Functional Gait Assessment (FGA) | before intensive therapy episode of care, an average of 4 weeks
  Assesses functional gait performance
Functional Gait Assessment (FGA) | after intensive therapy episode of care, an average of 4 weeks
  Assesses functional gait performance
Segmental Assessment of Trunk Control (SATCo) | before intensive therapy episode of care, an average of 4 weeks
  Assessment of trunk control
Segmental Assessment of Trunk Control (SATCo) | after intensive therapy episode of care, an average of 4 weeks
  Assessment of trunk control
Survey | after intensive therapy episode of care, an average of 4 weeks
  4 open-ended questions about caregiver/child experience with intensive therapy program

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Therapy Center--MU Healthcare, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No